CLINICAL TRIAL: NCT00621959
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating the Efficacy and Impact on Health-related Quality of Life of Levocetirizine 5 mg Once Daily Given for 2 Weeks in Subjects 18 yr of Age and Older With Seasonal Allergic Rhinitis
Brief Title: A Study Evaluating the Efficacy and Impact on Health-related Quality of Life of Levocetirizine in Adults With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00430
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: levocetirizine; Xyzal; Seasonal Allergic Rhinitis; total symptom score; quality of life
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo tablets once daily
  Interventions: Drug: placebo
- LCTZ (Experimental): 5 mg levocetirizine dihydrochloride tablet
  Interventions: Drug: levocetirizine dihydrochloride

INTERVENTIONS:
Drug: levocetirizine dihydrochloride — 5mg daily (oral tablet) for 14 days
  Other Names: Xyzal
  Arms: LCTZ
Drug: placebo — 0mg (matching oral tablet)for 14 days
  Arms: Placebo

SUMMARY:
The study objective is to investigate the efficacy of levocetirizine in reducing symptoms associated with seasonal allergic rhinitis and in improving rhinitis-related Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of SAR symptoms
* A positive skin prick test at least one grass allergen
* Moderate - severe SAR symptoms at baseline
* Women of childbearing potential must use a medically acceptable form of contraception
* 80% compliance on run in study medication and 80% compliance on completing the diary

Exclusion Criteria:

* The presence of any clinically significant comorbid disease which may interfere with the study assessments
* The presence of renal disease
* Pregnant or breastfeeding
* Subject is currently participating in another clinical trial
* Known hypersensitivity to piperazines or any of the excipients
* Intake of medications prohibited before the start of the trial
* Subjects who started or changed the dose of immunotherapy
* Rhinitis medicamentosa
* Subjects with a recent history (within the last 2 years) of drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (26):
- United States (26):
  - Scottsdale, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Huntington Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Mission Viejo, California
  - Albany, Georgia
  - Lilburn, Georgia
  - Savannah, Georgia
  - Owensboro, Kentucky
  - Metairie, Louisiana
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Katy, Texas
  - New Braunfels, Texas
  - Plano, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Waco, Texas

REFERENCES:
- [Derived] Segall N, Gawchik S, Georges G, Haeusler JM. Efficacy and safety of levocetirizine in improving symptoms and health-related quality of life in US adults with seasonal allergic rhinitis: a randomized, placebo-controlled study. Ann Allergy Asthma Immunol. 2010 Mar;104(3):259-67. doi: 10.1016/j.anai.2009.12.003. PMID 20377116
- [Derived] Mansfield LE, Hampel F, Haeusler JM, Georges G. Study of levocetirizine in seasonal allergic rhinitis. Curr Med Res Opin. 2010 Jun;26(6):1269-75. doi: 10.1185/03007991003745233. PMID 20350147
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- LCTZ: 5 mg levocetirizine dihydrochloride tablet once daily
Period: Overall Study
Arm/Group | Placebo | LCTZ
Started | 295 (In all 791 subjects have been screened and 596 have been randomized) | 301
Completed | 288 | 292
Not Completed | 7 | 9
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LCTZ | Total
Number analyzed (Participants) | 295 | 301 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.36 (11.05) | 37.02 (11.99) | 37.18 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 206 | 405
  Male | 96 | 95 | 191
Region of Enrollment [Number; unit: participants]
  United States | 295 | 301 | 596

OUTCOME MEASURES:

1. Primary Outcome: Mean 24-hour Reflective Total 5 Symptoms Score (T5SS)
Description: Total 5 Symptoms Score (T5SS) is the sum of rhinorrhea, sneezing, nasal congestion, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). The total score varies from 0 to 15.
Time Frame: Over the total treatment period (14 days)
Population: Number of participants from the Intent-To-Treat (ITT) population with available T5SS over the Total Treatment Period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | LCTZ
Number analyzed (Participants) | 294 | 299
points on a scale | 8.96 (2.96) | 8.77 (3.28)
Statistical Analysis 1: Comparison: Placebo vs LCTZ; The Null Hypothesis for the primary endpoint is expressed as follows: 'The mean 24-hr reflective T5SS over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.546, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean T5SS is considered as different between the two treatment groups; ANCOVA including treatment and center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.14, 95% CI [-0.59 to 0.31] — The difference presented is 'Levocetirizine 5 mg - Placebo'

2. Secondary Outcome: Change From Baseline in Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score
Description: The RQLQ is a validated instrument composed of 28 questions covering 7 dimensions of health. Each question is scored on a scale of 0 to 6 (in which 0 = not troubled and 6 = extremely troubled), and the mean value for each health dimension is calculated. Overall health-related quality of life is expressed as the mean of the seven dimension scores. The overall RQLQ score varies from 0 to 6.
Time Frame: Baseline and endpoint, defined as the last available post-baseline observation during the two-week treatment period (in days)
Population: Number of participants from the Intent-To-Treat (ITT) population with available overall RQLQ score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | LCTZ
Number analyzed (Participants) | 294 | 299
points on a scale | -1.07 (1.26) | -1.12 (1.25)
Statistical Analysis 1: Comparison: Placebo vs LCTZ; The Null Hypothesis is expressed as follows: 'The mean change from baseline in overall RQLQ score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.442, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in overall RQLQ score is considered as different between the two treatment groups; ANCOVA on the change from baseline in overall RQLQ score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.08, 95% CI [-0.27 to 0.12] — The difference presented is 'Levocetirizine 5 mg - Placebo'

ADVERSE EVENTS:
Arm/Group | Placebo | LCTZ
Serious Adverse Events (participants affected / at risk) | 2/295 | 0/301
Other Adverse Events (participants affected / at risk) | 30/295 | 29/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=295) | LCTZ (N=301)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=295) | LCTZ (N=301)
Fatigue (General disorders) | 5 | 9
Headache (Nervous system disorders) | 20 | 10
Somnolence (Nervous system disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.